CLINICAL TRIAL: NCT01185665
Title: Predicting Outcome of Transcutaneous Electrical Nerve Stimulator (TENS) in Failed Back Surgery Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Evenepoel Kristof (Unknown); De Rudder Marc (Unknown); Dokter Moens Maarten (primary investigator) (Unknown); Prof. dr. Cattrysse Eric (Unknown); Prof. Dr. D'Haens Jean (Unknown)
Responsible Party: Dr. Moens Maarten, UZ Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: vubmtmoensTENS
Record Dates: First submitted 2010-08-19; First posted 2010-08-20 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-08

CONDITIONS: Failed Back Surgery Syndrome
Keywords: FBSS
MeSH Terms: conditions — Failed Back Surgery Syndrome | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TENS (Active Comparator): FBSS patients treated with TENS
  Interventions: Device: TENS
- Sham-TENS (Placebo Comparator): patients treated with Sham-Tens
  Interventions: Device: Sham-TENS

INTERVENTIONS:
Device: TENS — Transcutaneous Electrical Nerve Stimulator
  Arms: TENS
Device: Sham-TENS — TENS without electrical output, from the outside not different from a normal TENS
  Arms: Sham-TENS

SUMMARY:
The study investigates the feasibility and efficacy of Transcutaneous Electrical Nerve Stimulator (TENS) in a subgroup of patients with neuropathic pain. Those patients are suffering of neuropathic pain at the lower back and leg after spinal surgery with a predominance of pain in the leg.

DETAILED DESCRIPTION:
Derived from folk tradition, the notion that rubbing the skin over a painful area relieves pain, found scientific support in the gate-control theory proposed by Melzack and Wall 1. Since then, electrical stimulations for pain relief have spread worldwide.

The most known technique is Transcutaneous Electrical Nerve Stimulator (TENS). Surface electrodes are placed over the lower back (paravertebral at level L1-L2) it and the stimulation is delivered at high frequency and low intensity (below pain threshold), to produce an intense activation of Ab afferents and to evoke paresthesiae that cover the painful area.

In the literature about TENS in neuropathic pain a few controlled trials (classes II-IV) were found 2-8. The most studies dealt with painful diabetic neuropathy were very-high-frequency stimulation of lower-limb muscles were found more efficacious than standard TENS and low-frequency TENS or acupuncture-like more efficacious than sham stimulations.

Studies dealing with peripheral mononeuropathies found standard TENS better than placebo.

One crossover, small-sample study (class III) in painful cervical radiculopathy found that standard TENS applied to the cervical back was better than placebo but a TENS with random frequency variation was superior7. For chronic back pain no benefit was found for TENS compared to TENS-sham using a VAS and other outcome measures, but benefit was found comparing exercise to no exercise (Class I)9. In another Class I study, TENS vs TENS-sham was studied in patients with multiple sclerosis (MS) and chronic low back pain. After correction for multiple comparisons, there were no significant differences in the VAS or the secondary measures10. Both studies were adequately powered to find at least a 20% difference in pain reduction by VAS between TENS and TENS-sham. But in other articles no benefit were found for chronic back pain treated with TENS11,12. Therefore a recent report of the Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology did not recommend TENS for the treatment of chronic low back pain due to lack of proven efficacy but TENS should be considered for the treatment of painful diabetic neuropathy 13

In our study design, we will investigate the feasibility and efficacy of TENS in a subgroup of patients with neuropathic pain. Those patients are suffering of neuropathic pain at the lower back and leg after spinal surgery with a predominance of pain in the leg.

ELIGIBILITY:
Inclusion Criteria:

Inclusions:

* Age male/female patient ≥ 18 years
* Patient diagnosed with Failed Back Surgery Syndrome with at least one prior spinal surgery
* Patient with low back pain and/or pain in at least one leg
* Pain intensity at baseline assessed by VAS > 5 (50%)

Exclusion Criteria:

Exclusions:

* Formerly treated with TENS
* Several unrelated sites of pain
* Cognitive impairment
* No help to replace electrodes
* Ongoing litigation
* Psychological intervention
* Language difficulties
* No informed consent
* Existing or planned pregnancy
* Age male/female patient <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility to use TENS devices in Failed Back Surgery Syndrome (FBSS) as a non-invasive method to treat neuropathic pain. | 1 year
  To evaluate the feasibility to use TENS devices in Failed Back Surgery Syndrome (FBSS) as a non-invasive method to treat neuropathic pain using pain scores, QOL scores and depression scores

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Moens, M.D., Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Vlaams Brabant, Belgium